CLINICAL TRIAL: NCT07378280
Title: A Randomized, Double-blinded, Placebo-controlled, Multi-center Study to Investigate the Effect of L. Lactis CKDB001 Administration on Liver Aminotransferases in Subjects With Nonalcoholic Fatty Liver Disease
Brief Title: Study to Investigate the Effect of L. Lactis CKDB001 Administration on Liver Aminotransferases in Subjects With NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Collaborators: Chong Kun Dang Bio (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CKDB001-01
Record Dates: First submitted 2024-10-20; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Non Alcoholic Fatty Liver Disease
Keywords: Non Alcoholic Fatty Liver; Probiotics; Gut-Liver Axis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The selected test subjects were randomly assigned to placebo and L. lactis CKDB001 group according to the order registered at visit 2 (week 0) after a 2-week run-in period, and treated with placebo for 12 weeks. After treatment, primary and secondary outcomes were analyzed.
  Interventions: Dietary Supplement: Placebo
- L. lactis CKDB001 (Experimental): The selected test subjects were randomly assigned to placebo and L. lactis CKDB001 group according to the order registered at visit 2 (week 0) after a 2-week run-in period, and treated with L. lactis CKDB001 (5.0E+09 CFU/day) for 12 weeks. After treatment, primary and secondary outcomes were analyzed.
  Interventions: Dietary Supplement: Probiotics (L. lactis CKDB001)

INTERVENTIONS:
Dietary Supplement: Probiotics (L. lactis CKDB001) — L. lactis CKDB001: Enteric coated capsule with L. lactis CKDB001, daily, 12 weeks
  Arms: L. lactis CKDB001
Dietary Supplement: Placebo — Placebo: Enteric coated capsule without any probiotics, daily, 12 weeks
  Arms: Placebo

SUMMARY:
A study for evaluating the safety and efficacy of L. lactis CKDB001 on liver aminotransferases in subjects with nonalcoholic fatty liver disease

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women aged 19 to 75 years at the time of written consent
* Voluntarily provided written consent after receiving sufficient explanation about the study
* ALT or AST levels exceed the upper limit of normal, but are five times or less than the upper limit

Exclusion Criteria:

* Pregnant or breastfeeding women
* Women of childbearing potential and men who are unable or unwilling to use appropriate contraception during the study period
* Individuals with a history of alcohol abuse or chronic alcohol consumption:

Daily alcohol consumption averaging over 30g/day (210g/week) for men or over 20g/day (140g/week) for women

* Individuals with viral or other liver diseases that could affect study results:
* Individuals with a history of or current drug abuse
* Individuals with a history of psychiatric disorders or current psychiatric conditions that may interfere with the study
* Individuals with a history of major gastrointestinal surgery (excluding appendectomy, but including gastric resection, gastrointestinal bypass, anastomosis, bariatric metabolic surgeries)
* Individuals with severe comorbidities that make them unsuitable for study participation (e.g., heart disease, kidney disease, malignancy, immunosuppression, etc.):
* Regular consumption of probiotics, prebiotics, synbiotics, or fermented milk within 4 weeks prior to screening (participation allowed if consumption ceases at least 1 month before study start)
* Regular consumption of medications, health supplements, or herbal remedies that may affect liver function or anti-inflammatory responses within 4 weeks prior to screening (participation allowed if consumption ceases at least 1 month before study start)
* Use of medications that may cause hepatic steatosis (e.g., amiodarone, tamoxifen, methotrexate, tetracycline, corticosteroids)
* Use of medications for treating non-alcoholic fatty liver disease (NAFLD) or steatohepatitis (NASH) within 3 months prior to screening (e.g., thiazolidinediones, vitamin E)
* Use of medications that may affect study results (e.g., antipyretic analgesics, NSAIDs, anti-tuberculosis drugs, antibiotics, anticonvulsants, choleretics, liver disease medications)
* Use of oral steroids, hormones, or drugs that may affect absorption, metabolism, or excretion of food within 4 weeks prior to screening (participation allowed if taking systemic steroids or thyroid hormones in stable doses for ≥3 months before screening)
* Use of hypoglycemic agents or lipid-lowering drugs (except insulin or thiazolidinediones) with stable doses for at least 3 months prior to screening
* Dietary or exercise therapies that may affect study within 3 months prior to screening
* Smokers consuming more than 20 cigarettes per day
* Allergies or digestive issues related to study food ingredients
* Weight loss exceeding 10% of previous body weight within 6 months prior to screening
* Participation in another clinical trial within 30 days prior to screening or not completing the required five-half-life period of investigational drug/food from a previous trial
* Any other individuals deemed unsuitable for the study by the investigator

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Changes in liver function parameters: AST (U/L), ALT (U/L) | From baseline to 12 weeks
  Change from baseline to 12 weeks in the specified liver function parameters will be assessed.

SECONDARY OUTCOMES:
Changes in liver function parameters: γ-GTP (U/L), ALP (U/L) | From baseline to 12 weeks
  Change from baseline to 12 weeks in the specified liver function parameters will be assessed.
Changes in bilirubin parameters: Total bilirubin (mg/dL), Direct bilirubin (mg/dL) | From baseline to 12 weeks
  Change from baseline to 12 weeks in the specified bilirubin parameters will be assessed.
Changes in protein parameters: Total protein (g/dL), Albumin (g/dL), Globulin (g/dL) | From baseline to 12 weeks
  Change from baseline to 12 weeks in the specified protein parameters will be assessed.
Changes in lipid parameters: Total cholesterol (mg/dL), LDL-C (mg/dL), HDL-C (mg/dL), Triglycerides (mg/dL) | From baseline to 12 weeks
  Change from baseline to 12 weeks in the specified lipid parameters will be assessed.
Changes in fasting plasma glucose levels (mg/dL) | From baseline to 12 weeks
  Change from baseline to 12 weeks in fasting plasma glucose levels will be assessed.
Changes in fasting serum insulin levels (μU/mL) | From baseline to 12 weeks
  Change from baseline to 12 weeks in fasting serum insulin levels will be assessed.
Changes in insulin resistance index: HOMA-IR | From baseline to 12 weeks
  Change from baseline to 12 weeks in the insulin resistance index (HOMA-IR) will be assessed.
Changes in inflammatory markers: TNF-α (pg/mL), IL-6 (pg/mL), IL-10 (pg/mL) | From baseline to 12 weeks
  Change from baseline to 12 weeks in the specified inflammatory cytokine markers will be assessed.
Changes in high-sensitivity C-reactive protein levels (mg/L) | From baseline to 12 weeks
  Change from baseline to 12 weeks in high-sensitivity C-reactive protein levels will be assessed.
Changes in Fatigue Severity Scale (FSS) | From baseline to 12 weeks
  Change from baseline to 12 weeks in Fatigue Severity Scale (FSS) score will be assessed. The FSS is a validated 9-item questionnaire with total scores ranging from 9 to 63, where higher scores indicate greater fatigue severity.
Changes in gut environment assessed by metagenomics and metabolomics | From baseline to 12 weeks
  Change from baseline to 12 weeks in gut environment will be assessed using metagenomic and metabolomic analyses.
Changes in body weight (kg) | From baseline to 12 weeks
  Change from baseline to 12 weeks in body weight will be assessed.
Changes in body mass index (kg/m²) | From baseline to 12 weeks
  Change from baseline to 12 weeks in body mass index will be assessed.
Changes in waist circumference (cm) | From baseline to 12 weeks
  Change from baseline to 12 weeks in waist circumference will be assessed.
Changes in hip circumference (cm) | From baseline to 12 weeks
  Change from baseline to 12 weeks in hip circumference will be assessed.
Changes in waist-to-hip ratio (WHR) | From baseline to 12 weeks
  Change from baseline to 12 weeks in waist-to-hip ratio will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Hallym University Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do, South Korea